CLINICAL TRIAL: NCT06316089
Title: An Intervention to Improve HIV Pre-exposure Prophylaxis Initiation, Adherence and Linkage to Care for Recently Incarcerated Men Who Inject Drugs.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Matthew Murphy, Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23DA054003 (NIH)
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Hiv; Substance Use Disorders
Keywords: HIV; Substance Use Disorders; Injection Drug Use; Incarceration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEPared For Release (Experimental): Intervention arm
  Interventions: Behavioral: PrEPared for Release
- Standard of Care (No Intervention): Control arm

INTERVENTIONS:
Behavioral: PrEPared for Release — A multilevel, behavioral and navigation intervention administered over two sessions to promote PrEP initiation, adherence and linkage to PrEP care in the community for incarcerated men with a history of injection drug use.
  Arms: PrEPared For Release

SUMMARY:
Pre-exposure prophylaxis (PrEP) is effective in preventing HIV infection among people who inject drugs (PWID) yet studies suggest that its use is low among this population which is particularly vulnerable to HIV infection. The criminal justice (CJ) system, at the intersection of increased risk of HIV infection and substance use, presents a unique opportunity to engage PWID in HIV prevention care that incudes PrEP. The study will characterize the facilitators and barriers to PrEP initiation, adherence and linkage to care among male PWID that are experiencing incarceration and develop the "PrEPare-for-Release" intervention to promote PrEP initiation, adherence and linkage to care upon release from incarceration into the community.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Incarcerated at the Rhode Island Department of Corrections
* Identifies as male
* Reports a history of injection drug use
* Meets CDC clinical criteria for PrEP use
* Able to provide written and verbal consent in either English or Spanish

Exclusion Criteria:

* Unable to provide written and/or verbal consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | Rapid, within 7 days
  Initiation of PrEP usage

SECONDARY OUTCOMES:
Adherence to PrEP | At least 30 days
  Appropriate use of PrEP postinitiation
Linkage to PrEP care in the community | Within 30 days post-incarceration
  Linkage to a community PrEP care provider for participants post-release from incarceration